CLINICAL TRIAL: NCT04082689
Title: Bowel And Bladder Function in Infant Toilet Training- a Randomized Intervention Study to Investigate the Efficacy of Assisted Infant Toilet Training on Preventing Functional Gastrointestinal and Urinary Tract Disorders up to 4 Years of Age
Brief Title: Bowel And Bladder Function in Infant Toilet Training
Acronym: BABITT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dalarna County Council, Sweden (Other)
Collaborators: Center for Clinical Research Dalarna, Sweden (Other); Örebro University, Sweden (Other); Göteborg University (Other)
Responsible Party: Principal Investigator, Barbro Hedin Skogman, Senior consultant at the Department of Paediatrics, Falun Hospital, Associate professor at Örebro Universitet, post-doctoral researcher at the Center for Clinical Research (CKF) Dalarna, Sweden, Dalarna County Council, Sweden
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: BABITT-01
Record Dates: First submitted 2019-06-12; First posted 2019-09-09 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Infantile Colic; Constipation - Functional; Bladder Dysfunction; Toilet Training
Keywords: Colic; Constipation; Bladder dysfunction; Toilet training
MeSH Terms: conditions — Colic; Constipation

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial (RCT) where one group of children who begin assisted infant toilet training at age 0-2 months (group A) is compared to a group of children who begin assisted infant toilet training at 10-11 months (group B).
Who Masked: Outcomes Assessor
Masking Description: The group allocation of the participating Children will be masked to the co-workers performing the ultrasound measurement of rectal diameter at 9 months and 4 years of age.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Assisted Infant Toilet Training-Group A (Active Comparator): Parents to Children randomized to group A will be instructed in how infant toilet training is performed by the investigators. They receive a book in Swedish concerning infant toilet training and a brief summary of the book made by the investigators. The parents are encouraged to begin infant toilet training as early as possible, 0-2 months of age
  The definition of adherence to the intervention is to perform at least one attempt a day of infant toilet training (without the requirement of a successful outcome) on at least 5 out of 7 days per week.
  Interventions: Behavioral: Assisted Infant Toilet Training
- Assisted Infant Toilet Training- Group B (Active Comparator): Parents to Children randomized to group B will be instructed in how infant toilet training is performed by the co-workers doing the ultrasound measure of rectal diameter at 9 months. They receive a book in Swedish concerning infant toilet training and a brief summary of it made by the investigators. They start infant toilet training at the age of 10-11 months.
  The definition of adherence to the intervention is to perform at least one attempt a day of infant toilet training (without the requirement of a successful outcome) on at least 5 out of 7 days per week.
  Interventions: Behavioral: Assisted Infant Toilet Training

INTERVENTIONS:
Behavioral: Assisted Infant Toilet Training — The parents learn to sensitively respond to the child's routines and signals of elimination needs.The child's ability to convey the need for bowel and bladder evacuation is enhanced through responsive interaction so that a kind of assisted dryness is developed. The infant is held "squatting" over a potty or basin, while older children sit on the potty.
  Other Names: Elimination Communication

SUMMARY:
The overall purpose is to assess whether assisted infant toilet training during the first year of life can prevent functional gastrointestinal and urinary tract disorders up to 4 year of age. Healthy Swedish children will be randomized to start assisted infant toilet training at 0-2 months of age or at 10-11 months of age.

The toilet training process will be described including mother-to-infant attachment and parental stress.

DETAILED DESCRIPTION:
The mastery of toilet training is an important developmental milestone for children and parents. The age at which children start toilet training has increased during the last decades in the Western world. 50 years ago most children were out of nappies by 1,5 years of age. Today, wearing nappies by 3-4 years of age is considered normal. Meanwhile an increase in functional gastrointestinal and urinary tract disorders and toileting problems is reported by health care professionals.

A randomized multicenter intervention study is conducted at Child Health Care Centers in Sweden to investigate whether assisted infant toilet training initiated during the first year of life can prevent functional bowel and bladder disorders.

ELIGIBILITY:
Inclusion Criteria:

* Full-term infant (born at gestational week 37+0 to 41+6)

Exclusion Criteria:

* Infants with malformations or disorders that may affect the gastrointestinal or urinary tract in any relevant way
* Infants born small for gestational age (SGA), < - 2 standard deviation
* Parents with insufficient understanding of the Swedish language
* Infants older than 2 months, 1 week and 6 days at inclusion

Max Age: 2 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 293 (Actual)
Dates: Start 2019-04-18 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Prevalence of functional constipation | Up to 9 months of age
  Functional constipation, measured with validated questionnaires according to the ROME IV criteria
Prevalence of infant dyschezia | Up to 9 months of age
  Infant dyschezia, measured with validated questionnaires according to the ROME IV criteria
Prevalence of infant colic | Up to 5 months of age
  Infant colic measured with validated questionnaires according to the ROME IV criteria, including a prospective 24h infant behavioral diary when infant colic is suspected

SECONDARY OUTCOMES:
Prevalence of functional constipation | Up to 4 years of age
  Functional constipation, measured with validated questionnaires according to the ROME IV criteria.
Prevalence of gastrointestinal symptoms | At 4 years of age
  Gastrointestinal symptoms, measured with Pediatric Quality of Life Inventory Gastrointestinal Symptoms Module (PedsQL Gastro)
Prevalence of stool toileting refusal | At 4 years of age
  Stool toileting refusal, measured with validated questionnaire
Prevalence of bladder dysfunction | Up to 4 years of age.
  Bladder dysfunction, measured with validated questionnaires according to International Childrens Continence Society (ICCS) definitions.

OTHER OUTCOMES:
Infant-to-mother attachment | Up to 9 months of age
  Infant-to-mother attachment, measured with Maternal Postnatal Attachment Scale (MPAS). It contains 19 issues, questions are scored 1-5. Total score is calculated by adding scores on all issues. Scale range for total score is 19-95. High score indicates higher mother-to-infant attachment.
Parental stress | Up to 2,5 years of age
  Parental stress, measured with Swedish Parental Stress Questionnaire (SPSQ). It contains 34 issues each scoring 1-5. Total score is calculated as an average on answers (1-5) on all issues. Scale range for total score is 34-170. High score indicates higher parental stress.

CONTACTS AND LOCATIONS:
Overall Officials: Barbro Hedin Skogman, assoc. prof., Study Director — Dalarna County Council, Sweden
Locations (6):
- Sweden (6):
  - Unicare vårdcentral Borlänge, Borlänge, Dalarna County
  - Vårdcentral Kvarnsveden, Borlänge, Dalarna County
  - Elsborgs Familjecentral, Falun, Dalarna County
  - Falu Vårdcentral, Falun, Dalarna County
  - Familjecentralen Bönan, Leksand, Dalarna County
  - Barnavårdscentral Mora, Mora, Dalarna County

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nilsson T, Leijon A, LoMartire R, De la Calle Dahlstedt S, Sillen U, Hellstrom AL, Skogman BH. Assisted infant toilet training and the prevalence of functional gastrointestinal disorders up to the age of 9 months: a randomised, controlled trial. Arch Dis Child. 2025 Nov 17:archdischild-2025-328792. doi: 10.1136/archdischild-2025-328792. Online ahead of print. PMID 41249012
- [Derived] Nilsson T, Leijon A, Sillen U, Hellstrom AL, Skogman BH. Bowel and bladder function in infant toilet training (BABITT) - protocol for a randomized, two-armed intervention study. BMC Pediatr. 2022 May 19;22(1):294. doi: 10.1186/s12887-022-03355-6. PMID 35590259

DOCUMENTS (2):
  • Study Protocol (2023-10-29): https://cdn.clinicaltrials.gov/large-docs/89/NCT04082689/Prot_007.pdf
  • Statistical Analysis Plan (2023-10-29): https://cdn.clinicaltrials.gov/large-docs/89/NCT04082689/SAP_008.pdf